CLINICAL TRIAL: NCT02374164
Title: A Phase 1, Open-Label, Single-Center, Randomized, 3-Way Crossover Study to Assess the Effect of Food on the Bioavailability of a Single Oral Dose of 80 mg Febuxostat Extended-Release Formulation and the Pharmacokinetics of a Single Oral Dose of 40 mg and 80 mg Febuxostat Extended-Release Formulation in Healthy Subjects
Brief Title: Food Effect Study of Febuxostat XR in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Febuxostat-XR-1009; U1111-1165-0441 (Registry Identifier: UTN (WHO))
Record Dates: First submitted 2015-02-22; First posted 2015-02-27 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Gout
Keywords: Drug therapy
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Sequence ABC (Experimental): Febuxostat extended release (XR) 80 mg, capsules, orally, once on Day 1 of Period 1 after a high-fat meal, followed by a 7-day washout period, followed by febuxostat XR 40 mg, capsules, orally, once on Day 1 of Period 2 after a 10-hour fast, followed by a 7-day washout period, followed by febuxostat XR 80, capsules, orally, once on Day 1 of Period 3 after a 10-hour fast.
  Interventions: Drug: Febuxostat XR
- Treatment Sequence BCA (Experimental): Febuxostat XR 40 mg, capsules, orally, once on Day 1 of Period 1 after a 10-hour fast, followed by a 7-day washout period, followed by febuxostat XR 80 mg, capsules, orally, once on Day 1 of Period 2 after a 10-hour fast, followed by a 7-day washout period, followed by Febuxostat XR 80 mg, capsules, orally, once on Day 1 of Period 3 after a high-fat meal.
  Interventions: Drug: Febuxostat XR
- Treatment Sequence CAB (Experimental): Febuxostat XR 80 mg, capsules, orally, once on Day 1 of Period 1 after a 10-hour fast, followed by a 7-day washout period, followed by febuxostat XR 80 mg, capsules, orally, once on Day 1 of Period 2 after a high-fat meal, followed by a 7-day washout period, followed by febuxostat XR 40 mg, capsules, orally, once on Day 1 of Period 3 after a 10-hour fast.
  Interventions: Drug: Febuxostat XR

INTERVENTIONS:
Drug: Febuxostat XR — Febuxostat XR capsules

SUMMARY:
The purpose of this study is to assess the effect of food on the bioavailability of febuxostat after a single oral dose of 80 mg febuxostat XR and to evaluate the pharmacokinetics (PK) of febuxostat after single oral doses of 40 and 80 mg febuxostat XR.

DETAILED DESCRIPTION:
The drug being tested in this study is called febuxostat extended- release (XR). This study is evaluating the effect of food on how febuxostat-XR moves throughout the body. This study will also look at the side effects and all safety results in people who took the study drug.

This 3-way crossover study will enroll approximately 36 participants. Eligible participants will be randomly (by chance) assigned to one of the 3 treatment sequences at 1:1:1 ratio. Sequence defines the order in which participants receive Regimens A (febuxostat XR 80 mg after a high fat meal), B (febuxostat XR 40 mg after fasting) and C (febuxostat XR 80 mg after fasting):

Sequence 1: A, B, C

Sequence 2: B, C, A

Sequence 3: C, A, B The dose in a period and the dose in the subsequent period will be separated by a minimum 7-day washout interval. This single-centre trial will be conducted in the United States.

Participants will make multiple visits to the clinic including three 4-day periods of confinement to the clinic, and will be contacted by telephone 30 days after last dose of study drug for a follow-up assessment.

.

ELIGIBILITY:
Inclusion Criteria:

1. Has an estimated glomerular filtration rate ≥90 mL/min.
2. Weighs at least 50 kg (110 pounds) and has a body mass index (BMI) from 18.0 to 30.0 kg/m^2, inclusive, at Screening.
3. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from the signing of the informed consent throughout the duration of the study and for 30 days after the last dose.
4. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after the last dose.
5. Able to attend all the visits scheduled in the study.
6. Willing to refrain from strenuous exercise from Day -1 until Study Exit (Day 3 of Period 3).

Exclusion Criteria:

1. Hypersensitivity to Febuxostat or to any of the components of the formulation.
2. Has received any investigational compound within 30 days prior to the first dose of study medication.
3. Has received febuxostat in a previous clinical study or as a therapeutic agent.
4. Has uncontrolled, clinically significant disease or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
5. Has a known hypersensitivity to any xanthine oxidase (XO) inhibitor, xanthine compounds, Febuxostat or any component of the formulation of Febuxostat tablets, or to caffeine.
6. Has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -1 of Period 1).
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
8. Is pregnant or lactating or intending to become pregnant before, during, or within 30 days post last dose; or intending to donate ova during such time period.
9. Intends to impregnate others or donate sperm during the course of this study or for 30 days post last dose.
10. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma, hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking febuxostat XR, or a similar drug in the same class, or a disease that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
11. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention [eg, cholecystectomy]).
12. Has a history of cancer, except basal cell carcinoma that has been in remission for at least 5 years prior to Day 1 of Period 1.
13. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or a known history of human immunodeficiency virus infection.
14. Has used nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, nicotine patch, or nicotine gum) within 28 days prior to Check-in (Day -1 of Period 1) or is unwilling to agree to abstain from nicotine-containing products. Cotinine test is positive at Screening or Check-in (Day 1 of Period 1).
15. Has poor peripheral venous access.
16. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis) or had a transfusion of any blood product within 30 days prior to Day 1 of Period 1.
17. Has a Screening abnormal (clinically significant) electrocardiogram (ECG).
18. Has abnormal Screening or Day -1 of Period 1 laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 x the upper limit of normal.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy participants took part in the study at 1 investigative site in the United States from 2 February 2015 to 19 April 2015.
Pre-assignment Details: Healthy participants were enrolled equally in 1 of 3 sequences which determined the order of treatment: Regimen A (febuxostat XR 80 mg after high fat meal), B (febuxostat XR 40 mg after fasting) and C (febuxostat XR 80 mg after fasting). Regimens included a single dose on Day 1 followed by a 7-day washout period prior to receiving the next regimen.
Period: Treatment Period 1
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 12 | 11 (One participant was Lost-to-Follow-Up prior to treatment A.) | 12
Completed | 12 | 11 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (8.37) | 35.0 (6.32) | 29.1 (5.35) | 31.8 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 7 | 19
  Male | 6 | 6 | 5 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 5 | 6 | 5 | 16
  Not Hispanic or Latino | 7 | 6 | 7 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 2 | 2 | 3 | 7
  White | 10 | 10 | 9 | 29
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36
Height [Mean (Standard Deviation); unit: cm] | 167.6 (8.27) | 168.8 (9.98) | 166.6 (12.35) | 167.6 (10.08)
Weight [Mean (Standard Deviation); unit: kg] | 73.95 (10.802) | 73.35 (8.867) | 69.10 (8.169) | 72.13 (9.335)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.21 (1.880) | 25.76 (2.321) | 25.03 (2.878) | 25.67 (2.376)
Female Reproductive Status [Number; unit: participants]
  N/A (Participant is Male) | 6 | 6 | 5 | 17
  Female of Childbearing Potential | 5 | 3 | 7 | 15
  Surgically Sterile | 1 | 3 | 0 | 4
Smoking Classification [Number; unit: participants]
  Has Never Smoked | 8 | 12 | 10 | 30
  Is a Current Smoker | 0 | 0 | 0 | 0
  Is an Ex-Smoker | 4 | 0 | 2 | 6
Alcohol Classification [Number; unit: participants]
  Has Never Drunk | 3 | 5 | 4 | 12
  Is a Current Drinker | 7 | 5 | 6 | 18
  Is an Ex-Drinker | 2 | 2 | 2 | 6
Xanthine/Caffeine Consumption [Number; unit: participants]
  Yes | 8 | 7 | 7 | 22
  No | 4 | 5 | 5 | 14
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min] — eGFR is calculated using the Cockcroft-Gault formula.
  mL/min
    Screening | 123.38 (22.449) | 125.41 (13.025) | 125.87 (15.280) | 124.88 (16.920)
    Check-in | 131.43 (25.231) | 132.71 (13.999) | 135.95 (19.147) | 133.36 (19.509)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Febuxostat XR 80 mg in Fed (Regimen A) and Fasted (Regimen C) States
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve. Participant blood samples were collected pre-dose and following a single oral dose.
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post dose
Population: Participants from the Pharmacokinetic population (PK), all participants who received study drug and had at least 1 measurable plasma concentration, who received a single dose of study drug in Regimen A and C.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- A: Febuxostat XR 80 mg (Fed): Febuxostat XR 80 mg, capsules, orally, once on Day 1 in any of the 3 treatment periods 30 minutes after starting to ingest a high-fat meal.
- C: Febuxostat XR 80 mg (Fasting): Febuxostat XR 80 mg, capsules, orally, once on Day 1 in any of the 3 treatment periods after a 10-hour fast.
Arm/Group | A: Febuxostat XR 80 mg (Fed) | C: Febuxostat XR 80 mg (Fasting)
Number analyzed (Participants) | 35 | 35
ng/mL | 1020.0000 (398.14171) | 1531.6286 (906.12813)
Statistical Analysis 1: Comparison: A: Febuxostat XR 80 mg (Fed) vs C: Febuxostat XR 80 mg (Fasting); Relative bioavailability of a single dose of Febuxostat XR 80 mg in the fasted and fed (high-fat meal) states; Test type: Superiority or Other; Point Estimate = 0.720, 90% CI 2-sided [0.612 to 0.847] — Ratio Fed/Fasted. Point estimate and 90% CI were obtained from the exponentiated results of analysis of the natural logarithm-transformed data. Bioequivalence was reached if the value was 0.80 to 1.25

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Febuxostat XR 40 mg (Regimen B) and Febuxostat XR 80 mg (Regimen C) in Fasted States
Description: as for outcome 1
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post dose
Population: Participants from the PK population, all participants who received study drug and had at least 1 measurable plasma concentration who received a single dose of study drug in Regimen B and C.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- B: Febuxostat XR 40 mg (Fasting): Febuxostat XR 40 mg, capsules, orally, once on Day 1 in any of the 3 treatment periods after a 10-hour fast.
Arm/Group | B: Febuxostat XR 40 mg (Fasting) | C: Febuxostat XR 80 mg (Fasting)
Number analyzed (Participants) | 36 | 36
ng/mL | 754.9167 (471.49630) | 1562.1389 (911.65824)

3. Primary Outcome: AUCt: Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Time of the Last Quantifiable Concentration for Febuxostat XR 80 mg in Fed (Regimen A) and Fasted (Regimen C) States
Description: AUCt is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration. Participant blood samples were collected pre-dose and following a single oral dose.
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post dose
Population: Participants from the PK population, all participants who received study drug and had at least 1 measurable plasma concentration, who received a single dose of study drug in Regimen A and C.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | A: Febuxostat XR 80 mg (Fed) | C: Febuxostat XR 80 mg (Fasting)
Number analyzed (Participants) | 35 | 35
ng*hr/mL | 7605.4147 (2086.85262) | 7687.1220 (2853.12475)

4. Primary Outcome: AUCt: Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Time of the Last Quantifiable Concentration for Febuxostat XR 40 mg (Regimen B) and Febuxostat XR 80 mg (Regimen C) in Fasted States
Description: AUCt is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUCt) Participant blood samples were collected pre-dose and following a single oral dose.
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post dose
Population: Participants from the PK population, all participants who received study drug and had at least 1 measurable plasma concentration, who received a single dose of study drug in Regimen B and C.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | B: Febuxostat XR 40 mg (Fasting) | C: Febuxostat XR 80 mg (Fasting)
Number analyzed (Participants) | 36 | 36
ng*hr/mL | 3646.2021 (1465.07275) | 7854.2007 (2985.41297)

5. Primary Outcome: AUCinf: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for Febuxostat XR 80 mg in Fed (Regimen A) and Fasted (Regimen C) States
Description: AUCinf is a measure of total plasma exposure to the drug from time zero extrapolated to infinity. Participant blood samples were collected pre-dose and following a single oral dose.
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | A: Febuxostat XR 80 mg (Fed) | C: Febuxostat XR 80 mg (Fasting)
Number analyzed (Participants) | 34 | 34
ng*hr/mL | 7816.0704 (2105.40456) | 8075.5899 (2826.48142)

6. Primary Outcome: AUCinf: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for Febuxostat XR 40 mg (Regimen B) and Febuxostate XR 80 mg (Regimen C) in Fasted States
Description: as for outcome 5
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | B: Febuxostat XR 40 mg (Fasting) | C: Febuxostat XR 80 mg (Fasting)
Number analyzed (Participants) | 35 | 35
ng*hr/mL | 3745.2837 (1452.71754) | 7970.7990 (2852.78221)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to 30 days after the last dose of study drug (approximately 58 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Set included all participants who received at least 1 dose of study drug.
Arm/Group | A: Febuxostat XR 80 mg (Fed) | B: Febuxostat XR 40 mg (Fasting) | C: Febuxostat XR 80 mg (Fasting)
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 1/35 | 3/36 | 2/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A: Febuxostat XR 80 mg (Fed) (N=35) | B: Febuxostat XR 40 mg (Fasting) (N=36) | C: Febuxostat XR 80 mg (Fasting) (N=36)
Nausea (Gastrointestinal disorders) | 0 | 2 | 1
Headache (Nervous system disorders) | 1 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.